CLINICAL TRIAL: NCT06996821
Title: Evaluation of Impacted or Included Maxillary Canines on Dentofacial Structures, and Airway and Nasal Fossa Dimensions
Acronym: Sinuses@Canine
Status: Completed | Type: Observational
Sponsor: JAVIER MONTERO (Other)
Responsible Party: Sponsor-Investigator, JAVIER MONTERO, Clinical Professor, University of Salamanca
Organization: University of Salamanca (Other)
Other Study IDs: 01/321; 01/321 (Other: Universidas Alfonso X El Sabio)
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: Impacted Canines; Maxillary Sinus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study retrospectively analyzed previously acquired CBCT images to evaluate specific anatomical features, such as [e.g., "maxillary sinus and nasal fossa volumes"]. No active patient participation or new clinical procedures is required; this information is used to measure sinus and fossa dimensions.

DETAILED DESCRIPTION:
The study analysed the CBCTs of patients, each assigned to one of three groups: control, unilateral canine impaction, or bilateral canine impaction. Each group was assigned by gender. Three values were analysed: maxillary sinuses left (MSL) and right (MSR), and sinuses with fossa MSNF measures in mm3.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral canine inclusion,
* young pacients between 10 and 23 years old.

Exclusion Criteria:

* pregnant women,
* major craniofacial deformities (such as cleft palate, severe asymmetric malocclusion, trauma or head & neck oncologic surgery),
* surgeries other than maxillomandibular advancement,
* patients with maxillary compression or syndromes
* any nasal or nasopharyngeal airway obstruction.
* skeletal, dental or dentoalveolar transversal or vertical issues

Ages: 10 Years to 23 Years | Sex: All
Age Groups: Child, Adult
Study Population: Orthodontic Department of Alfonxo X Sabio Masters' Clinics
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Different Volumes of Maxillary Sinuses and Nasal Airway Complex | November 2024 to February 2025
  Volume (in mm³) of the right maxillary sinus, left maxillary sinus, and combined nasal and maxillary sinus airway complex, measured using cone-beam computed tomography (CBCT) and Dolphin Imaging software. Measurements are performed in axial, coronal, and sagittal planes using standardized sensitivity and anatomical reference points.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Madrid, Spain